CLINICAL TRIAL: NCT00659477
Title: Comparison Safety and Efficacy of Basal Insulin Lantus® (Insulin Glargine) vs NPH Insulin in Combination With OADs in Patients With DMT2, Assessed by Continuous Glucose Monitoring System (CGMS). Multicentre, Prospective, Open- Label, Single Arm, Comparative Study in Patients Switched From NPH Insulin to Insulin Lantus®.
Brief Title: Comparison Safety and Efficacy of Basal Insulin Lantus® (Insulin Glargine) vs NPH Insulin in Combination With Oral Antidiabetic Drugs (OADs) in Patients With Diabetes Mellitus, Type 2 (DMT2)
Acronym: COBIN 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_02673; EudraCT #: 2007-003393-25
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin glargine — once daily
  Other Names: Lantus

SUMMARY:
Aim of the study is to compare two treatment regimens (insulin Lantus as basal insulin vs insulin NPH) plus oral antidiabetics in type 2 diabetic patients and confirm superiority of insulin glargine. Comparison is focused on: blood glucose (BG) variability of the two treatment regimens, quality of diabetes compensation (HbA1c, FBG/Fasting blood glucose), body weight development, dose of insulin and occurrence of symptomatic hypoglycaemia and other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2
* Patients treated NPH insulin with stable dosage of OADs (Oral antidiabetic drugs) for at least 2 months prior to study start and OADs treatment with metformin at least 1,7 g /day in combination with sulfonylurea or glinides.
* Patients must have a HbA1c range of >= 4,5% ( 6,2% DCCT/Diabetes Control and Complication Trials) and <= 8% ( 9,4 % DCCT/Diabetes Control and Complication Trials)
* Ability and willingness to perform continuous glucose monitoring system / CGMS (examination within the study)
* Written informed consent obtained prior to enrollment in the study
* Women are either not of childbearing potential or women of childbearing potential must not be pregnant and must use a reliable contraceptive measure for the duration of the study

Exclusion Criteria:

1. Fasting value C peptide <= 400 pmol/l
2. Active proliferative diabetic retinopathy, as defined by the application of photocoagulation or surgery, in the 6 months before study entry or any other unstable rapidly progressing retinopathy that may require photocoagulation or surgery during the study.
3. Pregnant women or women planning gravidity during clinical study protocol
4. Breast-feeding
5. History of hypersensitivity to the study drugs or to drugs with a similar chemical structure
6. Treatment with systemic corticosteroids in the 3 months prior to study entry and during study and other treatment, that can significantly have impression to glycaemia.
7. Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
8. Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major disease making implementation of the protocol or interpretation of the study results difficult
9. Impaired hepatic function as shown by Alamine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) greater than three times the upper limit of normal range at study entry
10. Impaired renal function as shown by serum creatinine >/= 133 micromol/L in men and >/= 124 micromol/L in women at study entry
11. History of drug or alcohol abuse in the last year
12. Mental condition causing the patient unable to understand the nature, scope and possible consequences of the study
13. Patient unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits and unlikelihood of completing the study
14. Use of insulin glargine outside the scope of the current SPC (Summary of Product Characteristics)

16. Patients included in other clinical studies

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The change in blood glucose variability | before start with insulin glargine treatment and at the end of the study

SECONDARY OUTCOMES:
Occurrence of adverse events | From signing of informed consent to the end of study
Development of diabetes compensation - fastig blood glucose and HbA1 | before starting therapy with Lantus and at the end of study
Development of weight of patients | Before starting Lantus vs at the end of the study
Comparison of dose of insulins NPH vs Lantus | Before starting Lantus and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Priborska, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Prague, Czechia

REFERENCES:
- [Derived] Zdarska DJ, Kvapil M, Rusavy Z, Krcma M, Broz J, Krivska B, Kadlecova P. Comparison of glucose variability assessed by a continuous glucose-monitoring system in patients with type 2 diabetes mellitus switched from NPH insulin to insulin glargine: the COBIN2 study. Wien Klin Wochenschr. 2014 Apr;126(7-8):228-37. doi: 10.1007/s00508-014-0508-6. Epub 2014 Feb 22. PMID 24563017